CLINICAL TRIAL: NCT04151160
Title: Using Point of Care Ultrasound to Measure Perioperative Edema in Infants With Congenital Heart Disease
Brief Title: Point of Care Ultrasound Measurements of Perioperative Edema in Infants With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: MuscleSound (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-1387
Record Dates: First submitted 2019-10-15; First posted 2019-11-05 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease; Edema; Fluid Overload
Keywords: MuscleSound
MeSH Terms: conditions — Heart Defects, Congenital; Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Case Subjects: Infants with hemodynamically significant congenital heart disease.
  Interventions: Diagnostic Test: Point of care ultrasound measurements
- Control Subjects: Healthy infants with no heart disease or non-hemodynamically significant congenital heart disease.
  Interventions: Diagnostic Test: Point of care ultrasound measurements

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound measurements — i. Ultrasound images will be obtained using a commercial, high frequency, linear Philips ultrasound probe attached to small, portable tablet. This tablet will have the capability of transferring the saved images to the secure MuscleSound cloud-based server.

SUMMARY:
Babies can be born with heart problems and sometimes need a heart surgery to fix the heart problem. Heart surgery can cause swelling from the build-up of extra fluid. Swelling can make it harder for babies to breath and has to be treated with medicine called diuretics. Swelling is hard to measure in babies, so it can be hard to know how much diuretic they need to treat the swelling. The investigators are looking for a better way to measure swelling in babies who have had heart surgery. Ultrasound uses sound waves to take pictures of the inside of the body. Ultrasound is used to take pictures of babies before they are born and to take pictures of their heart after they are born. New ultrasound software has been made from a company called MuscleSound that can quickly measure the amount of swelling in adults, usually in less than 2 minutes. This software has not yet been used to measure swelling in kids. This study plans to learn more about swelling in babies and will try to measure swelling in babies before and after heart surgery with the new ultrasound software. The study will also make the same measurements in babies who do not have heart disease to compare to babies having heart surgery.

DETAILED DESCRIPTION:
Congenital heart disease is the most common birth defect and occurs in ~8 per 1000 live births in the United States. Approximately 25% of these infants require surgery in the first year of life to repair or palliate their heart defect. Many cardiac surgeries require the use of cardiopulmonary bypass to maintain systemic blood flow and oxygen delivery during surgery. Cardiopulmonary bypass is not a natural process, and, as a result, contributes to post-operative physiologic derangements including ischemia-reperfusion injury, systemic inflammatory response, and subsequent fluid overload.

Fluid overload, in particular, is a common issue in children undergoing cardiac surgery, particularly in the immediate post-operative period. The rates of fluid overload following cardiothoracic surgery are high, reported between 31% and 100% in different studies depending on the method of assessment and the degree of fluid overload analyzed. Diaz et al demonstrated approximately 55% of children requiring mechanical ventilation or inotropic support in the intensive care unit developed fluid overload. Fluid overload is defined as a positive fluid balance and can occur extra or intravascularly. The buildup of excess extravascular fluid is also known as edema. The etiology of fluid overload and edema is multifactorial and includes fluid retention due neurohormonal pathway activation such as vasopressin and renin-angiotensin system, congestive heart failure, iatrogenic fluid administration, and capillary leak. Intravascular fluid overload can cause elevated central venous pressure, potentially leading to poor renal perfusion and subsequent acute kidney injury (AKI) while extravascular edema compromises abdominal and thoracic compliance and can make ventilation difficult. In the post-operative period, fluid overload has been associated with significant morbidity including AKI, longer mechanical ventilation dependence, prolonged length of stay, and increased mortality.

Unfortunately, management and treatment of fluid overload and edema are not standardized as it is currently difficult to accurately quantify the degree of fluid overload. Methods for monitoring fluid status include trending body weights, monitoring net fluid balance (intake versus output), trending central venous pressure, and physical exam findings. All of these current methods for monitoring fluid status can easily be confounded in the intensive care unit. A paucity of data exists regarding accurate methods of assessing edema in infants. Objective methods of evaluating fluid overload have been attempted, but are limited to measuring only intravascular volume, such as ultrasound of the jugular vein, or are difficult to apply clinically, such as skin bioelectric impedance. Additional research is needed to better understand and directly measure edema in infants.

Ultrasound of the skin is one possible method for quantifying extravascular fluid overload and edema through measurement of the thickness of skin and underlying subcutaneous layers. Ultrasound has previously been utilized in pediatric patients to diagnose skin and soft tissue infections, but there are no dedicated studies performed to solely measure edema. MuscleSound, an ultrasound technology company, has developed an automated software system to measure skin tissue structures, including edema, in adults. This technology has been studied in adults, however, it has not yet been trialed or validated in children. The ability to evaluate edema with a reliable, automated, non-invasive, bedside tool would provide objective measurements into a patient's fluid status. This tool would be of particular importance in infants with congenital heart disease who have many risk factors for fluid overload but whose fluid status can be difficult to appropriately assess.

ELIGIBILITY:
Case Subjects:

Inclusion Criteria:

* Age less than or equal to 12 months old at the time of enrollment
* Known hemodynamically significant congenital heart disease
* Undergoing surgery, with or without cardiopulmonary bypass, to repair or palliate their congenital heart defect

Exclusion Criteria:

* Known renal dysfunction
* Prematurity less than 36 weeks corrected gestational age

Control Subjects:

Inclusion Criteria:

* Age less than or equal to 12 months old at the time of enrollment
* No known heart disease OR presence of only non-hemodynamically significant congenital heart disease, including: tiny muscular ventricular septal defect, patent foramen ovale, peripheral pulmonary stenosis, normally functioning bicuspid aortic valve (no stenosis and no more than trivial insufficiency), and tiny patent ductus arteriosus

Exclusion Criteria:

* History of hemodynamically significant congenital heart disease
* History of surgery with general anesthesia
* Known renal dysfunction
* Prematurity less than 36 weeks corrected gestational age

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Case subjects: Infants with hemodynamically significant congenital heart disease.
  Control subjects: Healthy infants with no heart disease or non-hemodynamically significant congenital heart disease.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound Measurement of Edema | Up to Post-Op Day 5
  Depth (in millimeters) of edema from skin ultrasound measurements.

SECONDARY OUTCOMES:
Change in Daily Weight | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5
  Weight will be recorded in kilograms (kg)
Daily Fluid Balance (intake and output) | Up to Post-Op Day 5
  Hourly fluid intake and output will be measured in milliliters (mL)
CVP Measurements | Up to Post-Op Day 5
  Current central venous pressure (CVP) will be documented in millimeters of Mercury (mmHg) at the time of the each daily ultrasound
Documentation of edema | Up to Post-Op Day 5
  Presence of edema documented in the Electronic Medical Record (EMR)
Reports of pulmonary edema and/or pleural effusions on chest x-ray reports | Up to Post-Op Day 5
  Documentation of "pulmonary edema" and/or "pleural effusions". If pulmonary edema and/or pleural effusions are documented on chest x-ray, then this will be added to the study data collection form, including the documented severity (ranging from "minimal", "mild", "moderate", and "large")
Daily diuretic dose | Up to Post-Op Day 5
  Total amount of diuretics given in the post-operative period (and day prior to surgery).The diuretic dose over each 24 hour post-operative period (from post-operative day 0 up to post-operative day 5) will be divided by the subject's weight in kilograms leading to a total daily diuretic dose in "mcg/kg/day" or "mg/kg/day".
Daily positive pressure ventilation (invasive or non-invasive), | Up to Post-Op Day 5
  Documentation of mechanical ventilation, Continuous positive airway pressure (CPAP), Bilevel Positive Airway Pressure (BiPAP), Average volume-assured pressure support (AVAPS), and SiPAP. The number of days (rounding to the nearest half day) that a patient requires any of these forms of positive pressure ventilation will be documented.
Length of mechanical ventilation (hours), | Up to Post-Op Day 5
  Documentation of mechanical ventilation, CPAP, BiPAP, AVAPS, and SiPAP. The hours that a patient requires mechanical ventilation in the post-operative period will be calculated and documented
Intensive care unit length of stay (days) | Up to Post-Op Day 5
  The days spent in the intensive care unit in the post-operative period will be calculated and documented
Development of Acute Kidney Injury (AKI) using the Acute Kidney Injury Network (AKIN) scoring system | Up to Post-Op Day 5
  The AKIN scale will be used to assess the presence and severity of acute kidney injury (AKI). The AKIN is a classification/staging system of acute kidney injury developed by the Acute Kidney Injury Network which uses changes in serum creatinine (SCr) and urine output to assess AKI. Stages of acute kidney injury are defined as 1, 2, or 3, with 3 indicating the most severe AKI.
Post-operative mortality | Up to 30 days Post-Op
  Death during their hospitalization after surgery or within 30 days in the post-operative period

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Persson, MD, Principal Investigator — University of Colorado, Denver; Jesse Davidson, MD, Study Director — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Shuler CO, Black GB, Jerrell JM. Population-based treated prevalence of congenital heart disease in a pediatric cohort. Pediatr Cardiol. 2013 Mar;34(3):606-11. doi: 10.1007/s00246-012-0505-3. Epub 2012 Sep 14. PMID 22976198
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Raja SG, Dreyfus GD. Modulation of systemic inflammatory response after cardiac surgery. Asian Cardiovasc Thorac Ann. 2005 Dec;13(4):382-95. doi: 10.1177/021849230501300422. PMID 16304234
- [Background] Butler J, Rocker GM, Westaby S. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 1993 Feb;55(2):552-9. doi: 10.1016/0003-4975(93)91048-r. PMID 8431082
- [Background] Seguin J, Albright B, Vertullo L, Lai P, Dancea A, Bernier PL, Tchervenkov CI, Calaritis C, Drullinsky D, Gottesman R, Zappitelli M. Extent, risk factors, and outcome of fluid overload after pediatric heart surgery*. Crit Care Med. 2014 Dec;42(12):2591-9. doi: 10.1097/CCM.0000000000000517. PMID 25072753
- [Background] Hassinger AB, Wald EL, Goodman DM. Early postoperative fluid overload precedes acute kidney injury and is associated with higher morbidity in pediatric cardiac surgery patients. Pediatr Crit Care Med. 2014 Feb;15(2):131-8. doi: 10.1097/PCC.0000000000000043. PMID 24366508
- [Background] Diaz F, Benfield M, Brown L, Hayes L. Fluid overload and outcomes in critically ill children: A single center prospective cohort study. J Crit Care. 2017 Jun;39:209-213. doi: 10.1016/j.jcrc.2017.02.023. Epub 2017 Feb 16. PMID 28254390
- [Background] Wilder NS, Yu S, Donohue JE, Goldberg CS, Blatt NB. Fluid Overload Is Associated With Late Poor Outcomes in Neonates Following Cardiac Surgery. Pediatr Crit Care Med. 2016 May;17(5):420-7. doi: 10.1097/PCC.0000000000000715. PMID 27028790
- [Background] Sampaio TZ, O'Hearn K, Reddy D, Menon K. The Influence of Fluid Overload on the Length of Mechanical Ventilation in Pediatric Congenital Heart Surgery. Pediatr Cardiol. 2015 Dec;36(8):1692-9. doi: 10.1007/s00246-015-1219-0. Epub 2015 Jun 30. PMID 26123810
- [Background] Lex DJ, Toth R, Czobor NR, Alexander SI, Breuer T, Sapi E, Szatmari A, Szekely E, Gal J, Szekely A. Fluid Overload Is Associated With Higher Mortality and Morbidity in Pediatric Patients Undergoing Cardiac Surgery. Pediatr Crit Care Med. 2016 Apr;17(4):307-14. doi: 10.1097/PCC.0000000000000659. PMID 26914622
- [Background] Delpachitra MR, Namachivayam SP, Millar J, Delzoppo C, Butt WW. A Case-Control Analysis of Postoperative Fluid Balance and Mortality After Pediatric Cardiac Surgery. Pediatr Crit Care Med. 2017 Jul;18(7):614-622. doi: 10.1097/PCC.0000000000001170. PMID 28492405
- [Background] Lombel RM, Kommareddi M, Mottes T, Selewski DT, Han YY, Gipson DS, Collins KL, Heung M. Implications of different fluid overload definitions in pediatric stem cell transplant patients requiring continuous renal replacement therapy. Intensive Care Med. 2012 Apr;38(4):663-9. doi: 10.1007/s00134-012-2503-6. Epub 2012 Feb 11. PMID 22327560
- [Background] van Asperen Y, Brand PL, Bekhof J. Reliability of the fluid balance in neonates. Acta Paediatr. 2012 May;101(5):479-83. doi: 10.1111/j.1651-2227.2012.02591.x. Epub 2012 Jan 27. PMID 22220764
- [Background] Bontant T, Matrot B, Abdoul H, Aizenfisz S, Naudin J, Jones P, Dauger S. Assessing fluid balance in critically ill pediatric patients. Eur J Pediatr. 2015 Jan;174(1):133-7. doi: 10.1007/s00431-014-2372-9. Epub 2014 Jul 4. PMID 24990494
- [Background] Brooks ER, Fatallah-Shaykh SA, Langman CB, Wolf KM, Price HE. Bioelectric impedance predicts total body water, blood pressure, and heart rate during hemodialysis in children and adolescents. J Ren Nutr. 2008 May;18(3):304-11. doi: 10.1053/j.jrn.2007.11.008. PMID 18410888
- [Background] Avcil M, Kapci M, Dagli B, Omurlu IK, Ozluer E, Karaman K, Yilmaz A, Zencir C. Comparision of ultrasound-based methods of jugular vein and inferior vena cava for estimating central venous pressure. Int J Clin Exp Med. 2015 Jul 15;8(7):10586-94. eCollection 2015. PMID 26379848
- [Background] Deol GR, Collett N, Ashby A, Schmidt GA. Ultrasound accurately reflects the jugular venous examination but underestimates central venous pressure. Chest. 2011 Jan;139(1):95-100. doi: 10.1378/chest.10-1301. Epub 2010 Aug 26. PMID 20798190
- [Background] Nieman DC, Shanely RA, Zwetsloot KA, Meaney MP, Farris GE. Ultrasonic assessment of exercise-induced change in skeletal muscle glycogen content. BMC Sports Sci Med Rehabil. 2015 Apr 18;7:9. doi: 10.1186/s13102-015-0003-z. eCollection 2015. PMID 25905021
- [Background] Hill JC, Millan IS. Validation of musculoskeletal ultrasound to assess and quantify muscle glycogen content. A novel approach. Phys Sportsmed. 2014 Sep;42(3):45-52. doi: 10.3810/psm.2014.09.2075. PMID 25295766
- [Background] Millan IS, Hill J and Wischmeyer PE. Measurement of skeletal muscle glycogen status in critically ill patients: a new approach in critical care monitoring. Critical Care. 2015;19:S141.